CLINICAL TRIAL: NCT01486030
Title: Effect of Exercise Stress Testing on Peripheral Gene Expression Using Corus CAD Diagnostic Test (Age, Sex, Gene Expression Score ASGES).
Brief Title: Effect of Exercise Stress Testing on Peripheral Gene Expression Using Corus CAD (or ASGES) Diagnostic Test
Acronym: EXERCISE
Status: Completed | Type: Observational
Sponsor: CardioDx (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: CDX_000012; EXERCISE (Other: CardioDx)
Record Dates: First submitted 2011-10-17; First posted 2011-12-06 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Coronary Artery Disease; Angina Pectoris; Chest Pain; Cardiovascular Diseases; Coronary Heart Disease; CAD; CVD; CHD
Keywords: Atherosclerosis; Corus CAD; Age/Sex/Gene Expression Score; ASGES; Gene Expression; GES; CAD; CVD; CHD; Precision Medicine; Exercise Stress Test; Coronary Artery Disease; Angina Pectoris; Chest Pain; Cardiovascular Disease; Coronary Heart Disease; EXERCISE
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Chest Pain; Cardiovascular Diseases; Coronary Disease; Atherosclerosis; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — RNA PAXgene
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Diagnostic Test: Corus CAD (ASGES) — Age/Sex/Gene Expression Score - ASGES

SUMMARY:
This is a prospective, single-center study that aims to evaluate the acute and delayed effect of exercise stress testing on the peripheral gene expression (PGE) levels using a predefined gene set established in the Corus CAD (Age/Sex/Gene Expression score - ASGES) test in subject with known obstructive coronary artery disease (CAD) and in control subjects (without known CAD).

DETAILED DESCRIPTION:
This is a prospective, single-center study. This protocol is a pilot study to investigate the effects of "acute" exercise (by exercise stress testing; modified Bruce protocol) on peripheral gene expression (PGE) levels as measured by Corus CAD score (Age/Sex/Gene Expression score - ASGES). Subjects will have blood sampling at baseline, at peak exercise, within 30 to 60 minutes post-exercise, at 24-36 hours post-exercise. The study will be stratified by presence of CAD and gender. An equal number of subjects with known CAD and normal controls will be enrolled. Equally, an equal number of men and women will be included. A screening CBC and HgbA1c will be performed to ensure the subject meets the intended use instruction for Corus CAD (ASGES). Data collection will include presence or absence of ECG ischemia with testing, as well as heart rate and blood pressure response to exercise with other ECG and dynamic variables. There will be four blood samples taken per subject as shown in the figure below.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 45-75 years old
2. Able to perform an adequate exercise stress test
3. Subjects with no known CAD and subjects with known CAD subjects

Exclusion Criteria:

1. Known severe CAD that will be unsafe to exercise stress patient
2. Current MI or high-risk acute coronary syndrome (including high-risk unstable angina
3. NYHA class III or IV congestive heart failure
4. Severe regurgitant or stenotic cardiac valvular lesion
5. Severe left ventricular systolic dysfunction
6. Active systemic infection in the preceding 2 months or chronic infection (e.g. HIV, Hepatitis B or C, Tuberculosis)**.
7. Protocol-specified rheumatologic, autoimmune or hematologic conditions
8. Known or suspected diabetes mellitus or documented Hemoglobin A1C (A test for people with diabetes that monitors their average blood sugar levels over a period of two to three months) percent within last 6 months; presume normal HgbA1c (used as a standard tool to determine blood sugar control for patients with diabetes.) if none documented.
9. Total WBC 11,000/ul from a CBC drawn within 7 days of enrollment
10. Inadequate exercise stress test.
11. Recipient of any organ transplant
12. Immunosuppressive or immunomodulatory therapy including any dose of systemic corticosteroids in the preceding two months
13. Chemotherapy in the preceding year
14. Major surgery in the preceding 2 months
15. Blood or blood product transfusion in the preceding 2 months

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-diabetic subjects will be enrolled at the Department of Cardiology, Mayo Clinic, Florida. Enrollment will not be randomized. Subjects will be enrolled based on achieving an equal number of men and women, and known Coronary Artery Disease or CAD (prior history of ischemia by stress test or a coronary catheterization documenting greater than or equal to 50% stenosis in any vessels within 12 months prior to enrollment) and no known CAD (controls - prior of history of coronary catheterization documenting less than or equal to 15% stenosis in any vessels within 12 months prior to enrollment). Enrollment will be stratified as shown below:
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Age/Sex/Gene expression score (ASGES) difference between peak exercise and baseline | up to 1 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zapien, MS, Study Director — CardioDx
Locations (1):
- Mayo Clinic Research Unit, Jacksonville, Florida, United States